CLINICAL TRIAL: NCT00789048
Title: The Influence of "Operating Table Position Simulating Radiographs" on Acetabular Cup Angle During Primary Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Leonid Kandel, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cupangle-HMO-CTIL
Record Dates: First submitted 2008-11-09; First posted 2008-11-11 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2008-11

CONDITIONS: Hip Osteoarthritis
Keywords: hip; arthroplasty; radiograph
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — X-Rays

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgeon doesn't see (No Intervention): The surgeon doesn't see the radiograph prior to surgery
- Surgeon does see (Experimental): The surgeon can see the radiograph prior to surgery
  Interventions: Other: radiograph

INTERVENTIONS:
Other: radiograph — One radiograph with the patient lying on his contralateral side
  Arms: Surgeon does see

SUMMARY:
Goal of the research

1. To check the viability of "Operating Table Position Simulating Radiographs", while positioned on the contralateral side.
2. To determine whether knowledge about the angles displayed on this radiograph (pelvic tilt) influences the accurate positioning of the acetabular cup during the Total Hip Replacement procedure.

DETAILED DESCRIPTION:
Type of research:

A prospective study.

Population:

A power study has been calculated in order to define the sample size. The results indicated that the following sample size will suffice:

* Study group: 50 consecutive patients undergoing a primary total hip replacement procedure
* Control group: 50 consecutive patients undergoing a primary total hip replacement procedure

Inclusion criteria:

1. Age>18
2. Candidate for primary total hip replacement
3. Agrees to participate in the study

Exclusion criteria:

1. Patient doesn't agree to participate in the study

Protocol:

Patients included in the research group and in the control group will undergo an "Operating Table Position Simulating " radiograph of the pelvis. The radiograph will be done in the following manner: the patient will be potisioned on the non-operated side in such way that his pelvis is perpendicular to the table. The legs are flexed in 30 degrees at the hip joints and 30 degrees at the knees. The plate with a grid will be placed behind the pelvis in a device with notches (which can be used to measure the angles later). After the total hip replacement the patients will undergo an A-P radiograph of the hip joints while lying on the back with the hip joints bent to 30 degrees to overcome the forward tilt of the pelvis. All of the radiographs will be performed in the presence of an orthopedic surgeon.

The control group will be the first group of patients. Their radiographs will be stored in a standalone file with controlled access rather than the general PACS system. The file will be opened only when the study is over. The radiologist will control the file and be responsible for this stage.

The study group will be the next group of patients. In this group the radiographs will be saved in the general PACS system. The radiographs with measurement of the lateral inclination of the pelvis, while lying in an "Operating Table Position" will be shown to the chief surgeon on the day of surgery or one day prior to it.

Both chief surgeons will not know about the study until the end of it. At the end of the study, a comparison of both groups' acetabular cup angles will be done. The angles will be measured twice. The first measurement will be done by a senior orthopedic surgeon specializing in joint replacement operations. The second one will be done by a senior radiologist specialized in skeletal radiology. If a difference of 5 degrees or more is found between the two measurements, a third measurement will be done by a third examiner.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18
2. Candidate for primary total hip replacement
3. Agrees to participate in the study

Exclusion Criteria:

1. Patient doesn't agree to participate in the study
2. Dysplastic hip, Crowe>1
3. After previous hip surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
acetabular cup angle | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel